CLINICAL TRIAL: NCT06784193
Title: A Phase 1 First-in-Human, Open-Label, Multicenter Study of OP-3136 in Adult Participants With Advanced or Metastatic Solid Tumors
Brief Title: Phase 1 Study of OP-3136 in Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Olema Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OP-3136-101
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Advanced or Metastatic ER+ HER2- Breast Cancer (mBC); Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC); Advanced or Metastatic Castration-Resistant Prostate Cancer (mCRPC); Metastatic Breast Cancer; Fulvestrant; Palazestrant
Keywords: KAT6 Inhibitor; Histone Acetyltransferase (HAT) Inhibitor; Epigenetic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1A Dose Escalation monotherapy (Experimental)
  Interventions: Drug: OP-3136
- Part 1B Dose Escalation in combination with fulvestrant (Experimental)
  Interventions: Drug: OP-3136; Drug: Fulvestrant
- Part 1C Dose Escalation in combination with palazestrant (Experimental)
  Interventions: Drug: OP-3136; Drug: Palazestrant
- Part 2A Dose Expansion monotherapy - mBC (Experimental)
  Interventions: Drug: OP-3136
- Part 2A Dose Expansion monotherapy - mCRPC (Experimental)
  Interventions: Drug: OP-3136
- Part 2B Dose Expansion in combination with fulvestrant OR palazestrant-mBC @ RDE 1 (Experimental)
  Interventions: Drug: OP-3136; Drug: Fulvestrant; Drug: Palazestrant
- Part 2B Dose Expansion in combination with fulvestrant OR palazestrant-mBC @ RDE 2 (Experimental)
  Interventions: Drug: OP-3136; Drug: Fulvestrant; Drug: Palazestrant

INTERVENTIONS:
Drug: OP-3136 — Selective inhibitor of HAT enzymes KAT6A and KAT6B
Drug: Fulvestrant — Selective estrogen receptor degrader (SERD)
  Arms: Part 1B Dose Escalation in combination with fulvestrant; Part 2B Dose Expansion in combination with fulvestrant OR palazestrant-mBC @ RDE 1; Part 2B Dose Expansion in combination with fulvestrant OR palazestrant-mBC @ RDE 2
Drug: Palazestrant — Complete estrogen receptor antagonist (CERAN)
  Arms: Part 1C Dose Escalation in combination with palazestrant; Part 2B Dose Expansion in combination with fulvestrant OR palazestrant-mBC @ RDE 1; Part 2B Dose Expansion in combination with fulvestrant OR palazestrant-mBC @ RDE 2

SUMMARY:
This is a first-in-human, open-label, multicenter phase 1 study to evaluate safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of OP-3136, a lysine acetyltransferases 6A and 6B (KAT6A/B) inhibitor, as monotherapy and in combination with other anticancer agents in participants with advanced solid tumors.

This study consists of 2 parts: a dose escalation part (Part 1) and dose expansion part (Part 2).

DETAILED DESCRIPTION:
Part 1A (Dose Escalation for OP-3136 Monotherapy): This part of the study will evaluate the safety, tolerability, and PK in a range of doses of OP-3136, a lysine acetyltransferases 6A and 6B (KAT6A/B) inhibitor, administered orally once daily to participants with ER+ HER2- advanced or metastatic breast cancer (mBC), advanced or metastatic castration resistant prostate cancer (mCRPC), or advanced or metastatic non-small cell lung cancer (mNSCLC), and determine the maximum tolerated dose (MTD) and the recommended dose/regimen for expansion (RDE).

Part 1B (Dose Escalation for OP-3136 in Combination with Fulvestrant): This part of the study will evaluate the safety and PK of OP-3136 administered in combination with fulvestrant in participants with ER+ HER2- mBC, and determine MTD and RDE for this combination.

Part 1C (Dose Escalation for OP-3136 in Combination with Palazestrant): This part of the study will evaluate the safety and PK of OP-3136 administered in combination with palazestrant in participants with ER+ HER2- mBC, and determine MTD and RDE for this combination.

Part 2A (Dose Expansion for OP-3136 Monotherapy): This part will evaluate two expansion cohorts at the monotherapy RDE from part 1 in participants with ER+ HER2- mBC and participants with mCRPC.

Part 2B (Dose Expansion for OP-3136 in Combination with Fulvestrant OR Palazestrant): This part will evaluate the RDEs for OP-3136 in combination with fulvestrant from Part 1B OR the RDEs of OP-3136 in combination with palazestrant in an expansion cohort in participants with ER+ HER2- mBC.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with advanced or metastatic ER+HER2- breast cancer, mCRPC, or NSCLC (Part 1) or advanced or metastatic ER+HER2- BC or mCRPC (Part 2).
* Part 1A (Dose escalation for OP-3136 monotherapy): Participants must have a tumor that is unresectable or metastatic and for which life prolonging measures do not exist or available therapies are intolerable or no longer effective.
* Part 1B (Dose escalation for OP-3136 in combination with fulvestrant): Participants with advanced or metastatic ER+ HER2- breast cancer that have progressed on or after at least 1 prior line of treatment that included endocrine therapy and CDK 4/6 inhibitor in advanced or metastatic setting and must have received no more than 2 prior lines of endocrine therapy (one of which must be in combination with CDK4/6 inhibitor) and no more than 1 prior line of chemotherapy or an antibody-drug conjugate in the advanced or metastatic setting.
* Part 1C (Dose escalation for OP-3136 in combination with palazestrant): Participants with advanced or metastatic ER+ HER2- breast cancer that have progressed on or after at least 1 prior line of treatment that included endocrine therapy and CDK 4/6 inhibitor in advanced or metastatic setting and must have received no more than 2 prior lines of endocrine therapy (one of which must be in combination with CDK4/6 inhibitor) and no more than 1 prior line of chemotherapy or an antibody-drug conjugate in the advanced or metastatic setting.
* Part 2A (Dose Expansion in ER+ HER2- mBC for OP-3136 monotherapy): Participants must have received up to 3 prior lines of endocrine therapy (one of which must be in combination with CDK4/6 inhibitor) and up to 1 prior line of chemotherapy or an antibody-drug conjugate.
* Part 2A (Dose Expansion in mCRPC for OP-3136 monotherapy): Participants must have received up to 4 lines of prior systemic therapy for prostate cancer. Prior therapy must include treatment with an androgen receptor pathway inhibitor(s).
* Part 2B (Dose Expansion in ER+ HER2- mBC for OP-3136 in combination with fulvestrant OR Dose Expansion in ER+ HER2- mBC for OP-3136 in combination with palazestrant): Participants must have progressed on or after at least 1 prior line of treatment that included endocrine therapy and CDK 4/6 inhibitor in advanced or metastatic setting. Participants must have received no more than 2 prior lines of endocrine therapy in the advanced or metastatic setting and no more than 1 prior line of chemotherapy or an antibody-drug conjugate in the advanced or metastatic setting.

Key Exclusion Criteria:

* Prior therapy with KAT6A/B inhibitor in any treatment setting.
* Participants with advanced/metastatic, symptomatic, visceral spread, that are at risk of life-threatening complications in the short term.
* Known active or symptomatic central nervous system (CNS) metastases, carcinomatous meningitis, leptomeningeal disease, or a spinal cord compression that require CNS-specific treatment, or participants who did not demonstrate clinical and radiologic stability during the last 2 months prior to the first dose of study treatment or require or are currently on steroid therapy for CNS metastases.
* History of cerebral vascular disease, including transient ischemic attack, within 6 months prior to the first dose of study treatment.
* History of or ongoing impaired cardiac function or clinically significant cardiac disease within 6 months prior to the first dose of study treatment.

Note: Additional inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities in the Dose Escalation Arms | Up to 28 days
Incidence of adverse events and laboratory abnormalities | Up to 26 months

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to 26 months
Time to maximum concentration (Tmax) | Up to 26 months
Area under the curve from time zero to 24 hours (AUC0-24) | Up to 26 months
Overall Response Rate (ORR) | Up to 26 months
Duration of Response (DOR) | Up to 26 months
Clinical Benefit Rate (CBR) | Up to 26 months

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - Florida Cancer Specialists, Sarasota, Florida
  - University Medical Center - New Orleans, New Orleans, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - START - Midwest, Grand Rapids, Michigan
  - SCRI Oncology Partners, Nashville, Tennessee
  - START - San Antonio, San Antonio, Texas
  - START - Mountain Region, West Valley City, Utah
- Cancer Research South Australia, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Undecided